CLINICAL TRIAL: NCT05495854
Title: Pilot Feasibility and Non-inferiority Study of a Strategy for the Detection and Treatment of Helicobacter Pylori Infections in Primary Care Guided by a Non-invasive Technique for the Detection of Helicobacter Pylori Infection and Clarithromycin Resistance by PCR Real Time in the Stool
Brief Title: New Strategy for the Detection and Treatment of Helicobacter Pylori Infections in Primary Care Guided by a Non-invasive PCR in Stool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HEPYPRIM
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- National Health Authority (HAS) strategy control (No Intervention)
- new strategy experimental (Experimental)
  Interventions: Diagnostic Test: PCR test in the stool

INTERVENTIONS:
Diagnostic Test: PCR test in the stool — Patients randomized to the "new strategy" arm will receive a prescription for an Hp serology and a stool self-collection kit . Only the result of the PCR test in the stool will be considered for this arm. A positive test will determine Hp infection and the indication for treatment.
  Arms: new strategy experimental

SUMMARY:
In France, every year 1 million people are explored for Helicobacter pylori infection and 200,000 receive eradication treatment. Faced with the high prevalence of Hp resistance to antibiotics, the Haute Autorité de Santé (HAS) has recommended since 2017 a treatment strategy guided by the results of bacteriological tests (culture and antibiogram and / or PCR) carried out from gastric biopsies. Guided therapy is more effective, cheaper, and better tolerated than empiric therapy (it includes fewer antibiotics). But the guided treatment is not used despite the recommendations because of the invasive nature of the endoscopy, the difficulty of culture and the non-reimbursement of the PCR. A new non-invasive test by real-time PCR performed on the stools of patients makes it possible to detect the Hp infection and its sensitivity to clarithromycin and therefore to guide the treatment with excellent performance as we have been able to demonstrate during a study including 1200 patients (Pichon et al J Clin Microbiol 2020). These characteristics allow this test to be used in primary care but has to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Person over 18 years old
* Patient affiliated or beneficiary of a social security scheme.
* Informed consent signed by the patient after clear and fair information about the study
* Patient registered on the list of patients who signed a doctor's statement with the investigating doctor.
* Patient with an indication for research and treatment of an Hp infection according to HAS recommendations:

Suffering from (at least one) Chronic dyspepsia, Iron deficiency anemia without a found cause or resistant to iron supplementation, Vitamin B12 deficiency without a found cause, familial gastric cancer DCDS, Immunological thrombocytopenic purpura in adulthood, ATCD of peptic ulcers or precancerous lesions that have not been eradicated, Long-term consumption of NSAIDs, Long-term PPI consumption, or Patient who received Hp eradication treatment without eradication control. or Patient with risk factors for gastric cancer: person related to a patient who has had stomach cancer (parents, brothers / sisters, children); or Patient with a syndrome of predisposition to digestive cancers (Hereditary non-polyposis colorectal carcinoma cancer HNPCC / Lynch syndrome) or Patient who has had a partial gastrectomy or endoscopic treatment of gastric cancerous lesions or Patient with pre-neoplastic gastric lesions (severe atrophy and / or intestinal metaplasia, dysplasia).

or Patient who has already undergone an endoscopy with detection of Hp but without antibiotic sensitivity test (biopsy not addressed in bacteriology) and for whom we want to undergo a guided treatment

Exclusion Criteria:

* Patient not benefiting from a Social Security scheme or not benefiting from it through a third party.
* Patient benefiting from enhanced protection, namely minors, pregnant or breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection and finally patients in emergency situations.
* Pregnant or breastfeeding women, women of childbearing age who do not have effective contraception (hormonal / mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy ).

Exclusion criteria related to non-compliance with ambivalence:

* Allergy to amoxicillin (suspected or documented)
* Contraindication to eso-gastro-duodenal fibroscopy and biopsies
* Use of antibiotic within 15 days before enrolment
* Patient with an indication to perform an endoscopy of the upper digestive system in Emergency according to the criteria of "the European Panel on the Appropriateness of Gastrointestinal Endoscopy (EPAGE II)": upper gastrointestinal hemorrhage, acute deglobulization without digestive hemorrhage externalized, ingestion of caustics, acute dysphagia or ingestion of foreign bodies
* Participating another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-02-03 (Estimated); Study Completion 2024-02-03 (Estimated)

PRIMARY OUTCOMES:
Cure rate assessed by the result of a urea breath test carried out 6 weeks after the end of treatment (proof of Hp eradication) | up to 4 months

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Vincent HELIS, Frontenay-Rohan-Rohan
  - philippe BRAVIN, Jarnac-Champagne
  - Gwenaelle FARCY, La Mothe-Saint-Héray
  - Marie ROCHEPEAU, La Mothe-Saint-Héray
  - Claude SAPIN, La Roche-Posay
  - Lise BLANCHARD, Mignaloux-Beauvoir
  - ARCHAMBAULT Pierrick, Nueil-les-Aubiers
  - Marc CHABANNE, Pont Labbe Darnoult
  - Elodie POUPIN, Saint-Germain-de-Marencennes
  - Vincent JEDAT, Saint-Jean-d'Angély
  - Christophe BONNET, Tonnay-Charente
  - ANDRIEUX Marine, Vaux-sur-Mer
  - FRECHE Bernard, Vaux-sur-Mer